CLINICAL TRIAL: NCT03286140
Title: A Randomised Clinical Trial to Compare Early Versus Delayed Endovenous Treatment of Superficial Venous Reflux in Patients With Chronic Venous Ulceration
Brief Title: Early Venous Reflux Ablation Ulcer Trial
Acronym: EVRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Birmingham (Other); Universidad de Granada (Other); University of Manchester (Other); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13HH0722
Record Dates: First submitted 2017-09-04; First posted 2017-09-18 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Venous Leg Ulcer
Keywords: endovenous ablation
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: The EVRA ulcer trial is a pragmatic; multicentre randomised clinical trial with participants randomised1:1 to either:
  1. 'Standard' therapy consisting of multilayer elastic compression bandaging/ stockings with deferred treatment of superficial reflux (usually once the ulcer has healed)
  2. Early endovenous treatment of superficial venous reflux(within 2 weeks) in addition to standard therapy
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment of ulcer healing photos
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy arm (Active Comparator): Multilayer elastic compression bandaging/ stockings with deferred treatment of superficial reflux (usually once the ulcer has healed)
  Interventions: Procedure: Delayed endovenous intervention
- Early arm (Experimental): Early endovenous treatment of superficial venous reflux(within 2 weeks) in addition to standard compression therapy
  Interventions: Procedure: Early endovenous ablation

INTERVENTIONS:
Procedure: Early endovenous ablation
  Arms: Early arm
Procedure: Delayed endovenous intervention
  Arms: Standard therapy arm

SUMMARY:
The EVRA study evaluates the effects of early endovenous ablation on ulcer healing in patients with chronic venous ulceration. Half the patients are randomised to receive early endovenous ablation (within 2 weeks) and half to standard care

DETAILED DESCRIPTION:
A large number of patients (around 1% of the adult population) suffer from an ulcer (break in the skin surface) near the ankle. In most people, such an injury should heal up within a week or two. However, when there is an underlying problem with the skin, ulcers do not heal and may result in longstanding (chronic), painful, smelly and embarrassing wounds. The ulcers are often due to varicose veins in the legs, which can cause skin breakdown and ulcer formation. To get the ulcer to heal, the current best treatment is to wear a tight compression bandage with multiple layers, with which about 60% of these ulcers will heal within 24 weeks. There is evidence that treatment of the varicose veins by surgery will prevent the ulcer from returning after it has healed. Recent studies have suggested that newer techniques of treating varicose veins, such as injecting a medicine into the varicose vein (sclerotherapy) or treating the vein with heat ablation to seal it (using laser or radiofrequency), in an outpatient setting may help the ulcers to heal more quickly and (like surgery) reduce the chance of the ulcer coming back. These techniques can be carried out in the outpatient setting and are much better tolerated by patients in comparison to surgery. The aim of this study is to see whether early treatment of varicose veins using sclerotherapy or heat ablation helps with healing.

ELIGIBILITY:
Inclusion Criteria:

* Current leg ulceration of greater than 6 weeks, but less than 6 months duration
* Able to give informed consent to participate in the study after reading the patient information documentation
* Patient age > 18 years
* Ankle Brachial Pressure Index (ABPI) ≥ 0.8
* Superficial venous disease on colour duplex assessment deemed to be significant enough to warrant ablation by the treating clinician (either primary or recurrent venous reflux)

Exclusion Criteria:

* Presence of deep venous occlusive disease or other conditions precluding superficial venous intervention (at the discretion of local research team)
* Patients who are unable to tolerate any multilayer compression bandaging / stockings will be excluded. However, concordance with compression therapy can be variable for patients at different times. Patients who are generally compliant with compression, but unable to tolerate the bandages for short periods will still be eligible to inclusion. A period of non-compliance with compression bandages will not be considered a protocol violation, but a normal variation within the spectrum of 'standard therapy'.
* Inability of the patient to receive prompt endovenous intervention by recruiting centre
* Pregnancy (female participants of reproductive age will be eligible for inclusion in the study, subject to a negative pregnancy test prior to randomisation)
* Leg ulcer of non-venous aetiology (as assessed by responsible clinician)
* Patient deemed to require skin grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Stansby, Study Chair — Newcastle University; Julie Brittenden, Study Chair — University of Glasgow
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At completion of the study, data will be shared in accordance with the NIHR HTA guidance on study outputs as per the research contract between the secretary of state for health research and Imperial College London. Only anonymised data will be shared under the terms of the consent forms.
  Data and associated documentation will be available to users only under a data-sharing agreement that provides for the following:
  1. A commitment to using the data only for research purposes and not to identify any individual participant;
  2. A commitment to securing the data using appropriate computer technology;
  3. A commitment to destroying or returning the data after analyses are completed. All requests are dealt with on a case-by-case basis. Any request should be submitted to the corresponding author who will then review with the Trial Management Group and sponsor. A record of all access to data will be maintained by the Imperial College Archive team.

REFERENCES:
- [Result] Gohel MS, Mora MSc J, Szigeti M, Epstein DM, Heatley F, Bradbury A, Bulbulia R, Cullum N, Nyamekye I, Poskitt KR, Renton S, Warwick J, Davies AH; Early Venous Reflux Ablation Trial Group. Long-term Clinical and Cost-effectiveness of Early Endovenous Ablation in Venous Ulceration: A Randomized Clinical Trial. JAMA Surg. 2020 Dec 1;155(12):1113-1121. doi: 10.1001/jamasurg.2020.3845. PMID 32965493
- [Result] Gohel MS, Heatley F, Liu X, Bradbury A, Bulbulia R, Cullum N, Epstein DM, Nyamekye I, Poskitt KR, Renton S, Warwick J, Davies AH. Early versus deferred endovenous ablation of superficial venous reflux in patients with venous ulceration: the EVRA RCT. Health Technol Assess. 2019 May;23(24):1-96. doi: 10.3310/hta23240. PMID 31140402
- See also: Trial website — https://www.imperial.ac.uk/department-surgery-cancer/research/surgery/clinical-trials/evra/

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Therapy Arm: Multilayer elastic compression bandaging/ stockings with deferred treatment of superficial reflux (usually once the ulcer has healed)
  Delayed endovenous intervention
- Early Arm: Early endovenous treatment of superficial venous reflux(within 2 weeks) in addition to standard compression therapy
  Early endovenous ablation
Period: Overall Study
Arm/Group | Standard Therapy Arm | Early Arm
Started | 226 | 224
6-week Follow-up | 224 | 223
6-month Follow-up | 215 | 213
12-month Follow-up | 203 | 204
Completed | 211 | 208
Not Completed | 15 | 16
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Lost to Follow-up | 5 | 10
Not completed — Failure to comply | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy Arm | Early Arm | Total
Number analyzed (Participants) | 226 | 224 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (14) | 67 (15.5) | 68 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 97 | 203
  Male | 120 | 127 | 247
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 208 | 206 | 414
  Mixed | 0 | 1 | 1
  Asian | 12 | 11 | 23
  Black | 5 | 3 | 8
  Other | 1 | 3 | 4
Weight (kg) [Mean (Standard Deviation); unit: kg] | 88.8 (24.1) | 89.5 (25.6) | 89.1 (24.9)
Height (cm) [Mean (Standard Deviation); unit: cm] | 170.5 (10.8) | 171.9 (11.1) | 171.2 (11.0)
BMI (kg/m2 ) [Mean (Standard Deviation); unit: kg/m2] | 30.4 (7.4) | 30.1 (7.8) | 30.3 (7.6)
Smoking [Count of Participants; unit: Participants]
  Current | 19 | 23 | 42
  Former | 101 | 86 | 187
  Never | 106 | 115 | 221
Previous ulcer [Number; unit: participants]
  Yes | 117 | 118 | 235
  No | 108 | 106 | 214
  Not completed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Ulcer Healing From Date of Randomisation to Date of Healing up to 365 Days
Description: For the purposes of this study, ulcer healing is defined as complete re-epithelialisation of all ulceration on the randomised (reference) leg in the absence of a scab (eschar) with no dressing required.
Time Frame: time from date of randomisation to date of healing up to 365 days
Population: For the purposes of this study, ulcer healing is defined as complete re-epithelialisation of all ulceration on the randomised (reference) leg in the absence of a scab (eschar) with no dressing required.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 226 | 224
days | 82 [69 to 92] | 56 [49 to 66]

2. Secondary Outcome: Percentage of Participants With Ulcer Healing
Description: Healing rate will be reported at 24 weeks using the percentage of participants with a healed ulcer
Time Frame: 24 weeks & time to ulcer healing up to 365 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 226 | 224
percentage of participants | 76.3 [70.5 to 81.5] | 85.6 [80.6 to 89.8]

3. Secondary Outcome: Ulcer Recurrence / Ulcer Free Time
Description: Will be calculated up to 1 year for each study arm and with the extension, up to 5 years (median approximately 3.7 years). This will allow a very practical and easily understood assessment of the clinical difference between the 2 arms of the study. This will also allow comparison with other studies that have reported this outcome. In order to facilitate accurate calculation of reoccurrence / ulcer free time, clinical follow up will be continued after ulcer healing up to 1 year after randomisation.
Time Frame: Up to 12 months (and with the extension, up to 5 years (median approximately 3.7 years))
Population: All participants with a healed ulcer within 1 year post-randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 194 | 210
Participants | 32 | 24

4. Secondary Outcome: Quality Of Life Questionnaire up to 365 Days
Description: Disease specific (AVVQ) quality of life
  The Aberdeen Varicose Vein Questionnaire (AVVQ) is a validated patient-reported disease-specific health questionnaire to assess quality of life in patients with varicose veins. The AVVQ comprises a diagram on which patients draw on their varicose veins and a questionnaire with 12 questions, half of which require a response for each leg. The scores range from 0 to 100 (no effect to severe effect).
Time Frame: 6 weeks post randomisation, 6 months, 12 months
Population: Missing data at follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 170 | 176
score on a scale
  6-week AVVQ | 41.2 (9.3) | 39.4 (10.2)
  6-month AVVQ: number analyzed (Participants) | 140 | 139
  6-month AVVQ | 39.5 (10.3) | 34.6 (9.4)
  12-month AVVQ: number analyzed (Participants) | 130 | 127
  12-month AVVQ | 34.3 (10.4) | 32.4 (8.3)

5. Secondary Outcome: Generic (SF-36) Quality of Life Assessment
Description: Generic (SF-36) quality of life assessment
  The Short Form questionnaire-36 items (SF-36) is a generic quality-of-life tool used to determine people's physical and mental health. It has been validated in many patient groups, including those with varicose veins. The physical domain measures physical functioning, physical role limitations, body pain and general health, whereas the mental dimension measures vitality, social functioning, mental health role limitations and general mental health. Two separate scores are produced (separate physical/mental component summary scores), in addition to the eight separate domain scores. Each score is measured on a scale of 0 to 100 (worst to best). Scores represent the percentage of total possible score achieved.
Time Frame: 6 weeks post randomisation, 6 months, 12 months
Population: SF-36 general health score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 207 | 212
score on a scale
  6-week SF-36 | 45.6 (9.2) | 45.7 (9.1)
  6-month SF-36: number analyzed (Participants) | 193 | 187
  6-month SF-36 | 44.5 (10.1) | 44.9 (9.8)
  12-month SF-36: number analyzed (Participants) | 181 | 183
  12-month SF-36 | 45.1 (10) | 45.3 (10)

6. Secondary Outcome: EuroQol-5 Dimensions (EQ-5D)
Description: The EuroQol-5 Dimensions (EQ-5D) is a widely recognised, generic tool to measure health outcomes and has been validated in a variety of patient groups, including those with venous leg ulcers. The EQ-5D questionnaire comprises two sections; the first assesses the participant's mobility, self-care, ability to perform usual activities, pain/discomfort and anxiety/depression levels, and the second records the participant's self-rated health on a vertical score of 0 to 100.
Time Frame: 6 weeks post randomisation, 6 months, 12 months
Population: EQ-5D health score Scores on the EuroQol Group 5-Dimension 5-Level questionnaire (EQ-5D-5L) health scale (a visual-analogue scale) range from 0 to 100, with higher scores indicating better health. Score on the EQ-5D-5L health index range from 0 to 1, with higher scores indicating better health. The EQ-5D-5L health index was calculated with the value set for England
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 205 | 212
score on a scale
  6-week EQ-5D | 71.1 (18.7) | 72.7 (18.6)
  6-month EQ-5D: number analyzed (Participants) | 193 | 185
  6-month EQ-5D | 71.4 (19.6) | 74.1 (15.8)
  12-month EQ-5D: number analyzed (Participants) | 184 | 183
  12-month EQ-5D | 73.7 (17.4) | 74.8 (16.9)

7. Secondary Outcome: Health Economic Assessment
Description: A within-RCT cost effectiveness analysis will be carried out based on the data collected in the trial, Resource use items in hospital and community care related to the treatment of venous ulceration or complications will be recorded for each patient at each follow-up. Resource use will be multiplied by UK unit costs obtained from published literature, HRG costs, and manufacturers' list prices to calculate overall costs. A standard tariff will be applied for each bandage change. Utilities (QALYs) will be calculated from the EQ-5D questionnaire administered to patients
Time Frame: Baseline, 6 weeks, 6 months, 12 months
Population: As randomised, less early withdrawals
Measure: Mean (Standard Deviation); unit: Costs (pounds) at one year
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 211 | 208
Costs (pounds) at one year | 2516 (3242) | 2514 (2770)

8. Secondary Outcome: Clinical Success - Presence of Residual / Recurrent Reflux in the Veins
Description: The presence of residual / recurrent varicose veins remaining on the venous duplex. Any reflux detected by the vascular scientists (as per local scanning policies) is recorded as presence of residual reflux and therefore considered incomplete clinical success. No presence of residual reflux is considered clinical success. (Clinical-Etiology-Anatomy-Pathophysiology) ranges from C0 which means absolutely no venous disease that can be seen or felt in the legs to C6 which means an open and active venous leg ulcer. For this outcome measure: Healed venous leg ulcer (C5), Active venous leg ulcer (C6).
Time Frame: at 6 weeks
Population: CEAP classification
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 226 | 225
Participants
  CEAP 5 | 1 | 1
  CEAP 6 | 225 | 224

9. Secondary Outcome: Clinical Success - VCSS
Description: The Venous Clinical Severity Score (VCSS) is a component of the Venous Severity Scoring System designed in 2000 by an ad hoc American Venous Forum committee consensus, in order to compliment the CEAP classification and quantify the severity of disease and subsequent improvement or decline. The VCSS has 10 components (pain, varicose veins, venous oedema, skin pigmentation, inflammation, induration, compression used and active ulcer, duration, number and size), each with four categories assigned values of 0-3. The overall scores can range from 0 (lowest severity) to 30 (highest severity).
Time Frame: at 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 226 | 224
score on a scale | 12.6 (4.4) | 10.5 (4.7)

10. Secondary Outcome: Clinical Success - Complications
Description: Number of complications related to the endovenous intervention
Time Frame: up to 12 months
Measure: Number; unit: participants
Arm/Group | Standard Therapy Arm | Early Arm
Number analyzed (Participants) | 226 | 224
participants | 24 | 28

ADVERSE EVENTS:
Time Frame: AEs collected over 12-months
Description: The research nurses collected data regarding the occurrence of all SAEs via the monthly telephone calls, clinic or surgery notes, and hospital admission records. These were reported to the ICTU via the web-based data capture system within 24 hours of the nurses becoming aware of the event and reviewed by the chief investigator.
Arm/Group | Standard Therapy Arm | Early Arm
All-Cause Mortality (participants affected / at risk) | 4/226 | 3/224
Serious Adverse Events (participants affected / at risk) | 51/226 | 40/224
Other Adverse Events (participants affected / at risk) | 83/226 | 67/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy Arm (N=226) | Early Arm (N=224)
Hospitalisation Required (General disorders) | 50 | 38
Other (General disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy Arm (N=226) | Early Arm (N=224)
New ulcer (Vascular disorders) | 83 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT03286140/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03286140/SAP_001.pdf